CLINICAL TRIAL: NCT07396623
Title: Validation of the French Versions of the PHQ-4 Anxiety and Depression Scale and the PC-PTSD-5 Post-Traumatic Stress Disorder Screening Scale
Brief Title: Validation of French PHQ-4 and PC-PTSD-5 Screening Scales
Acronym: DEPSYSTAGE
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP250750
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Mental Illness
Keywords: Post-Traumatic Stress Disorder; Depression; Anxiety; Screening tool
MeSH Terms: conditions — Mental Disorders; Stress Disorders, Post-Traumatic; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 554 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Mental illness is a major public health issue. It affects one in five people, represents the largest expense for health insurance (14%), is the leading cause of years lived with disability, and suicide is the main cause of death among people aged 15 to 35. Depression affects 15 to 20% of individuals at some point in their lives. Trauma-related disorders affect 4.6% of people, including 1- 2% with post-traumatic stress disorder (PTSD).

Screening for mental health problems in primary care is crucial. It enables doctors to provide early treatment, reduces the need for emergency care, and decreases both the number and duration of hospital stays. However, general practitioners and other non-mental health professionals often report lacking the time, training, and tools to conduct such screenings. Fortunately, brief and validated screening tools exist in English: The PHQ-4 (Patient Health Questionnaire-4) for anxiety and depression, and the PC-PTSD-5 (Primary Care PTSD Screen for DSM-5) for PTSD. So far, no French versions of these tools have been validated.

DETAILED DESCRIPTION:
A target of 10 patients per item of the tested scales was set. The PHQ-4 includes four items and the PC-PTSD-5 includes five items, corresponding to required sample sizes of 40 and 50 patients, respectively. Although the same patient sample completes both scales, these sample sizes were combined to account for potential loss to follow-up and to optimize statistical power, resulting in a total inclusion target of 90 patients.

Descriptive analyses of sociodemographic and clinical characteristics will be conducted for all included patients. Quantitative variables will be summarized using means and standard deviations, and qualitative variables using frequencies and percentages.

To address the primary objective, convergent validity will be assessed using Pearson's correlation coefficients between scores obtained on the tested scales (PHQ-4 and PC-PTSD-5) and those obtained on their respective gold standard instruments (PHQ-9, GAD-7, and PCL-5). Convergent validity will also be examined by inclusion center through comparison of correlation coefficients across centers.

Secondary objectives will be addressed through:

* Exploratory factor analysis to examine the dimensional structure of each scale and to compare it with that of the corresponding gold standard.
* Assessment of internal consistency using Cronbach's alpha coefficient. Test-retest reliability will be evaluated using the intraclass correlation coefficient on a subsample of at least 20 participants, depending on the final total sample size, who will complete the PHQ-4 and PC-PTSD-5 scales twice.
* Evaluation of diagnostic performance by calculating sensitivity and specificity for each scale among patients undergoing a psychiatric diagnostic assessment, with receiver operating characteristic (ROC) curves generated for each scale.
* Assessment of feasibility based on the time required to complete both scales.

All statistical tests will be two-sided and considered statistically significant at an alpha level of 0.05.

No statistical imputation methods will be used for the management of missing data.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years,
* Outpatient or hospitalized for any health-related reason,
* Oral and written proficiency in French,
* Patient informed and willing to participate in the study,
* Patient with health insurance coverage

Exclusion Criteria:

* Individuals under legal protection measures (guardianship, conservatorship, or legal supervision),
* Other factors preventing obtaining non-opposition or conducting the research, such as: limited French proficiency, hearing impairment, or significant cognitive disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will involve adult patients, regardless of sex, who present for consultation.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2026-01-26 (Actual); Primary Completion 2027-08-15 (Estimated); Study Completion 2027-08-15 (Estimated)

PRIMARY OUTCOMES:
Assess the validity of the French version of the PHQ-4 (Patient Health Questionnaire-4 ) scale | 14 days
  This scale is used for the screening of anxiety and depression. The scale will be scored.
  Score ranging from 0 to 12, corresponding to four levels of psychological distress:
  * None: 0-2
  * Mild: 3-5
  * Moderate: 6-8
  * Severe: 9-12 Patients will complete this scale at Visit 1 and Visit 2.
Assess the validity of the French version of the PC-TDSD-5 (Primary Care PTSD Screen for DSM-5) scale | 14 days
  Scale assessing whether the patient has experienced unusually or particularly frightening, horrible, or traumatic events. Examples include:
  * A serious accident or fire
  * Physical or sexual assault, or sexual abuse
  * An earthquake or flood
  * War
  * Witnessing a person being killed or seriously injured
  * The death of a close person by homicide or suicide Total score = sum of "YES" responses to questions 1 through 5. Patients will complete this scale at Visit 1 and Visit 2.

SECONDARY OUTCOMES:
Assess the feasibility of this screening tool during the first evaluation visit. | At Visit 1 (at inclusion)
  The time required for the patient to complete each scale (individually) will be timed and recorded (without informing the patient in order to avoid potential stress).

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Avicenne, Bobigny, France

IPD SHARING:
Plan to Share IPD: No